CLINICAL TRIAL: NCT05446987
Title: Effect of Position Change and Back Massage Versus Early Ambulation on Post Transfemoral Coronary Angiography Complications
Brief Title: Position Change and Back Massage Versus Early Ambulation on Post Transfemoral Coronary Angiography Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Suad Elsaman, Assistant professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Transfemoral Complication
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Catheter Complications; Ambulation Difficulty; Bleeding; Back Pain; Oozing; Hematoma
Keywords: coronary angiography; Complications; Early ambulation; Position; Transfemoral; Back massage
MeSH Terms: conditions — Mobility Limitation; Hemorrhage; Back Pain; Hematoma | interventions — Early Ambulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Position change and back massage group (Experimental): The patients received changing of position every two hours as follows in the same order: supine position with a head angle of 15°, semi-fowler position with a head angle of 30°, lateral right or left position with a head angle of 15°. Also, the patients received a simple stroke of lower back massage for 5 minutes every 2 hours
  Interventions: Other: Position change and back massage
- Early ambulation (Experimental): The patient are allowed to ambulate after 3 hours of complete bed rest in the supine position with a zero head of bed elevation angle.
  Interventions: Other: Early ambulation

INTERVENTIONS:
Other: Position change and back massage — Changing the patient's position every two hours as follows in the same order: supine position with a head angle of 15°, semi-fowler position with a head angle of 30°, lateral right or left position with a head angle of 15°. Also, the researcher applied a simple stroke of lower back massage for 5 minutes every 2 hours
  Arms: Position change and back massage group
Other: Early ambulation — The patient ambulated after 3 hours of complete bed rest in the supine position with a zero head of bed elevation angle
  Arms: Early ambulation

SUMMARY:
The study aimed to assess the effect of position change and back massage versus early ambulation on post transfemoral coronary angiography complications.

DETAILED DESCRIPTION:
Post transfemoral coronary angiography (TFCA) may be associated with complications such as oozing, bleeding, ecchymosis, hematoma, and back pain. As a result, nursing practice must be geared toward enhancing patient safety post-transfemoral coronary angiography procedure. This study aimed to assess the effect of position change and back massage versus early ambulation on post transfemoral coronary angiography complications. A quasi-experimental research design was used to conduct this study at the Coronary Care Unit of the selected university hospital in Egypt. A convenience sample of 185 patients undergoing transfemoral coronary angiography was included in the study during the first 6 hours post-transfemoral coronary angiography and randomly assigned to two groups: 92 patients received position change and back massage (PCBM group), and 93 patients underwent early ambulation after the first 3 hours post-transfemoral coronary angiography (EA group). The used tool was "Post Transfemoral Coronary Angiography Complication Assessment".

ELIGIBILITY:
Inclusion Criteria:

* Mean arterial blood pressure ≥70 mmHg.
* Heart rate ≥ 60 b/m.
* Manual compression closure technique on the access site
* Partial thromboplastin time < 90 seconds.
* Prothrombin time <16 seconds).
* No anticoagulant therapy within 24 hours before the cardiac catheterization procedure.

Exclusion Criteria:

* Patients who had a history of previous coronary stents.
* chronic pain,
* chronic obstructive pulmonary disease.
* Renal failure,
* Hypercoagulable conditions such as protein C.
* Cardiopulmonary resuscitation during angiography.
* Femoral artery ruptures during angiography.
* Chest pain with new electrocardiograph change.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Oozing and bleeding scale | After six hours post transfemoral coronary angiography
  It was designed to measure any leakage of blood from the puncture site. It classified oozing and bleeding according to the surface area of the dressing soaked with blood to three items: (1) No bleeding or oozing (dry dressing), (2) Oozing (surface area < 2cm 2), (3) Bleeding (surface area ≥2cm 2).
  The researcher rated vascular complications on a dichotomous scale (Yes/No). The "Yes" response indicated the presence of complications and was given a score of one. On the other hand, the "No" response indicated the absence of complications and received a score of zero.
Ecchymosis and hematoma formation scale | After six hours post transfemoral coronary angiography
  It was designed to measure ecchymosis and hematoma size. It classified ecchymosis and hematoma according to the surface area of blood collection under the skin into three items: (1) No ecchymosis or hematoma (no blood collection), (2) Ecchymosis (surface area <2cm2), (3) Hematoma (surface area ≥ 2cm2). The researcher rated vascular complications on a dichotomous scale (Yes/No). The "Yes" response indicated the presence of complications and was given a score of one. On the other hand, the "No" response indicated the absence of complications and received a score of zero.
Numeric rating scale | After six hours post transfemoral coronary angiography
  The scale was used to assess the lower back pain intensity. It is a four-point numerical rating scale: no pain (0), mild pain (1-3), moderate pain (4-7), severe pain (8-10).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria University, Study Chair — Faculty of Nursing, Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau KW, Tan A, Koh TH, Koo CC, Quek S, Ng A, Johan A. Early ambulation following diagnostic 7-French cardiac catheterization: a prospective randomized trial. Cathet Cardiovasc Diagn. 1993 Jan;28(1):34-8. doi: 10.1002/ccd.1810280107. PMID 8416329
- [Background] Kim K, Won S, Kim J, Lee E, Kim K, Park S. Meta-analysis of complication as a risk factor for early ambulation after percutaneous coronary intervention. Eur J Cardiovasc Nurs. 2013 Oct;12(5):429-36. doi: 10.1177/1474515112462519. Epub 2012 Oct 17. PMID 23076977
- [Background] Steffenino G, Dellavalle A, Ribichini F, Russo P, Conte L, Dutto S, Giachello G, Lice G, Tomatis M, Uslenghi E. Ambulation three hours after elective cardiac catheterisation through the femoral artery. Heart. 1996 May;75(5):477-80. doi: 10.1136/hrt.75.5.477. PMID 8665340
- [Background] Wood RA, Lewis BK, Harber DR, Kovack PJ, Bates ER, Stomel RJ. Early ambulation following 6 French diagnostic left heart catheterization: a prospective randomized trial. Cathet Cardiovasc Diagn. 1997 Sep;42(1):8-10. doi: 10.1002/(sici)1097-0304(199709)42:13.0.co;2-8. PMID 9286529